CLINICAL TRIAL: NCT04812873
Title: The Prevalence of ID (Iron Deficiency) & IDA (Iron Deficiency Anemia) in Korean Patients With Heart Failure
Brief Title: Registry Study of ID & IDA in Korean Patients With Heart Failure
Acronym: HFRegistry
Status: Completed | Type: Observational
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JWP-FER-401
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum Ferritin, Hb, Iron, TSAT BNP(or NT-proBNP), RDW, platelet, WBC, neutrophil count, lymphocyte count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of Iron Deficiency and Iron Deficiency Anemia in Korean HF patient

DETAILED DESCRIPTION:
Epidemiological study to assess The prevalence of ID (Iron Deficiency) & IDA (Iron Deficiency Anemia) in Korean patients with heart failure

ELIGIBILITY:
Inclusion Criteria:

* more than 19 years old
* Informed Consent Form
* Hear Failure criteria as belows

  * Heart Failure Sign(more than 1 Sx such as fatigue, dyspnea, ankle swelling)

    * Heart Failure Symptom(more than 1 among Jugular venous pressure (JVP) elevation, pulmonary crackle, peripheral edema) ③ Lung congestion or edema at chest X-ray ④ Objective findings of structural or functional cardiac abnormality(more than abnormality level of BNP or NT-proBNP, abnormality of echocardiography )

Exclusion Criteria:

* Not applicable

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Korean patients with heart failure
Sampling Method: Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The Prevalence of Iron Deficiency | 1 day
  serum ferritin < 100 ㎍/L or serum ferritin 100-299 ㎍/L and TSAT* < 20%
The Prevalence of Iron Deficiency Anemia | 1 day
  include Iron Deficiency criteria & Male: Hb < 13 g/dL, Female Hb < 12 g/dL

SECONDARY OUTCOMES:
Current Anemia treatment | 1 day
  Number of Participants take Anemia Medication

CONTACTS AND LOCATIONS:
Overall Officials: SOOJIN JUN, Study Director — JWPharmaceuticals
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JJ, Yoon M, Cho HW, Lee SE, Choi JO, Yoo BS, Kang SM, Choi DJ. Iron Deficiency in Korean Patients With Heart Failure. J Korean Med Sci. 2023 Jun 12;38(23):e177. doi: 10.3346/jkms.2023.38.e177. PMID 37309696